CLINICAL TRIAL: NCT07000747
Title: Molecular and Cellular Basis of Severe Forms of Dengue in Sickle Cell Patients
Acronym: DREPADENGUE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH3_2023/09; 2019-A03033-54 (Other: ANSM Frech Human Health Organisation)
Record Dates: First submitted 2025-05-21; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Dengue (Virus); Fever, Sandfly; Sickle Cell Disease
Keywords: extracellular vesicles; blood immune cells; Dengue virus
MeSH Terms: conditions — Dengue; Virus Diseases; Fever; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — one blood collection will be realized during the annual follow up visit of the patients and during the screening visit for the controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients SS Group: Fifty SS patients
- Patients SC: Fifty SC patients
- Control group AA: Patients without hemoglobin disease

SUMMARY:
Dengue virus (DENV) belongs to the genus of Flavivirus transmitted by the mosquito Aedes aegypti and is responsible for an infectious disease associated with different forms and severities such as dengue hemorrhagic fever or shock syndrome. Several recent reports have shown that sickle cell patients exhibited an increased risk of developing severe forms of dengue episodes compared to non-sickle cell subjects. Furthermore, among major sickle cell syndromes, these studies suggest that SC patients are at the highest risk of death during these infectious episodes although this sickle cell syndrome is generally associated with a more moderate expression of sickle cell disease. However, the mechanisms involved remain unknown to date.

The aim of the present study is to identify the molecular and cellular basis of this increased severity of dengue in SC patients. We hypothesize an exacerbation during DENV infection of the inflammatory response in SC patients compared to SS patients.

DETAILED DESCRIPTION:
More precisely, the objective is to determine and compare the different cellular and molecular inflammatory mediators between SS and SC patients at baseline, and to study DENV-induced activation of various blood figurative elements isolated from uninfected sickle cell patients in vitro.

Given the essential role of immune cells in the DENV cycle and in the innate and adaptive immune responses of the host, understanding the changes induced by viral infection in Peripheral Blood Mononuclear Cells (PBMC) and Monocyte-Derived Dendritic Cells (MDDC) remains a priority. The effect of DENV or DENV-Associated Molecular Patterns (PAMPs) will therefore be studied in vitro on purified cells from SC and SS patients.

The impact of MicroParticles (MPs), known to be involved in the pathogenesis of severe dengue forms and in sickle cell disease, will also be evaluated on two cell types: endothelial cells and neutrophils, the latter exhibiting exacerbated activation and production of Neutrophil Extracellular Traps (NETs).

Considering the influence of mosquito saliva components on the pathogenesis of arboviruses (including DENV) in vertebrate hosts through the amplification of inflammatory responses, a comparative analysis of cellular and molecular inflammatory mediators released following exposure of blood cells from SS and SC patients to DENV and Aedes aegypti saliva will be conducted in vitro.

Lastly, the differential blood profiles of SS and SC patients will be assessed for their impact on the vector competence of Aedes aegypti mosquitoes in transmitting DENV.

ELIGIBILITY:
Inclusion Criteria:

* patients with SS or SC SCD or controls with hemoglobin AA
* diagnosis of SCD performed by electrophoresis or HPLC in a reference laboratory for hemoglobinopathies
* patients older than 6 years and younger than 25 at inclusion
* clinically in a steady state at inclusion (without complication during the last month and without transfusion in the three last months)
* patients followed up for SCD at the sickle cell center of Guadeloupe (University hospital of Guadeloupe, Pointe-à-Pitre)
* patients or legal representatives of minors who will provide written informed consent in accordance with the Declaration of Helsinki
* patients affiliated to national social security
* the control group (AA subjects) will be recruited among volunteers recruited by posters

Exclusion Criteria:

* patients with SS or SC SCD or controls with hemoglobin AA
* diagnosis of SCD performed by electrophoresis or HPLC in a reference laboratory for hemoglobinopathies
* patients older than 6 years and younger than 25 at inclusion
* clinically in a steady state at inclusion (without complication during the last month and without transfusion in the three last months)
* patients followed up for SCD at the sickle cell center of Guadeloupe (University hospital of Guadeloupe, Pointe-à-Pitre)
* patients or legal representatives of minors who will provide written informed consent in accordance with the Declaration of Helsinki
* patients affiliated to national social security
* the control group (AA subjects) will be recruited among volunteers recruited by posters

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients from 6 to 25 years, with sicke cell disease in a steady state at inclusion
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Lymphocyte subpopulations measured by flow cytometry at steady-state | baseline
  Comparison of circulating lymphocyte subpopulations in terms of activation and expression of markers of inflammation (cytokines, microparticles) and neutrophil proteome of SS and SC sickle cell patients at steady-state.

SECONDARY OUTCOMES:
activation status of immune cells induced by DENV | baseline
  Quantification and comparison of activation state of immune cells (PBMC/monocytes) isolated from SS and SC sickle cell patients induced in vitro by DENV and/or DENV PAMPS (such as NS1 viral protein) in the presence or absence of mosquito saliva
Comparative Analysis of NET Formation Induced by Sickle Cell-Derived Microparticles With or Without Mosquito Saliva | baseline
  Comparison of the induction properties of Neutrophil Extracellular Traps (NETs) in vitro by microparticles isolated from SS and SC patients in the presence or absence of mosquito saliva
Impact of SS and SC Blood Profiles on Aedes aegypti Biting Behavior and Dengue Virus Transmission | baseline
  Evaluation of the influence of SS and SC blood profiles on the biting behavior of Aedes aegypti and its ability to transmit DENV.

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Etienne-Julan, MD PhD, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- Chu de La Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No